CLINICAL TRIAL: NCT05895435
Title: THE EFFECT OF RADIOFREQUENCY ON POSTMENOPAUSAL ADIPOSE TISSUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Adel Elasyed Darahem, effect of radiofrequancy on postmenopausal adipose tissue, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: the effect of radiofrequancy
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Show Positive Effect of Radiofrequancy on Postmenopausal Adipose Tissue
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first group (Experimental): Group (A) (Control Group):
  It will be consisted of 30 patients who will receive aerobic exercise and diet for 8 successive weeks 2 sessions per week.
  Interventions: Other: aerobic exercise
- second group (Experimental): Group (B) (Study Group):
  It will be consisted of 30 patients who will receive aerobic exercise and diet and radiofrequency for 8 successive weeks 2 sessions per week.
  Interventions: Device: radiofrequancy; Other: aerobic exercise

INTERVENTIONS:
Device: radiofrequancy — * Power of device: 150 W
  * Duration of the session: 40 minutes
  * Frequency: 2 sessions per week for 8 week.
  * Heating temperature: According to patient tolerance.
  Arms: second group
Other: aerobic exercise — The program include five minutes for warming-up in the form of range of motion and stretching exercises, thirty minutes of walking on treadmill with high speed (60-70% of maximum heart rate) and five minutes of cooling down (on treadmill with low speed and without inclination

SUMMARY:
* Menopause is associated with a redistribution of adipose tissue towards central adiposity, known to cause insulin resistance. It was found that menopause was associated with changes in adipose tissue phenotype related to metabolic dysfunction. In subcutaneous adipose tissue (SAT)
* The radiofrequency uses high-frequency electromagnetic waves to produce heat at the cutaneous and the subcutaneous levels. The mechanism of action, through the vibration of water molecules, transforms the electromagnetic energy into thermal. The heat generated by conversion occurs under 30 kHz to 300 MHz, and the most frequently used frequency is set between 0.5 and 1.5 MHz. The RF mechanism of fat reduction occurs by the generation of thermal stimulation of adipocyte metabolism, occurring through enzymatic degradation by lipase-mediated triglycerides, apoptosis, and adipocyte rupture and the objective of study to show the positive effect of radiofrequancy on postmenopausal adipose tissue

DETAILED DESCRIPTION:
About 90% of menopausal women experience some amount of weight gain. It is a natural and common aspect of getting older. It occurs because the body mass increases, as a result of fat deposits. However, weight gain associated with menopause typically involves increased amounts of fat around the abdomen. On an average, women gain between 8-10 kilogram between the ages of 45 and 55, the stage in life when menopause occurs. This extra weight generally does not evenly distribute itself throughout a woman's body. The weight tends instead to accumulate around the abdomen or thighs (Singh et al., 2013).

Postmenopausal women are usually troubled by increasing weight and waist circumference caused by obesity and android fat redistribution it is mostly attributed to estrogen depletion though other factors such as chronological aging and decline in physical activity play a significant role. The deleterious health consequences of obesity and visceral fat deposition after menopause encompass a variety of problems; from dyslipidemia and metabolic syndrome to increased risk of cardiovascular disease (CVD), osteoporosis, malignancies and mortality (Stachowiak et al., 2015) This emphasizes the need of effective methods for treating central adiposity in post-menopausal woman. No prior studies have investigated the effect of radiofrequency on adipose tissue. So this may add a new physical therapy method for treating this problem.

ELIGIBILITY:
Inclusion Criteria:

* 1-Their ages will be ranged from 45 to 60 years 2- BMI > 25 kg/m² and < 35 kg/m². 3- Waist circumference more than 88cm

Exclusion Criteria:

* 1-Cancer. 2-Renal failure 3-tumors 4-Hepatic diseases 5-skin disease that prevent the use of radiofrequancy

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-18 (Estimated)

PRIMARY OUTCOMES:
total cholestrol and HDL and LDL and triglycerides and VLDL by blood analysis | 8 week
  measure before and after tratement programm

SECONDARY OUTCOMES:
waist circumferance using tape measurment | 8 week
  measure before and after tratement
body mass index | 8 week
  measure before and after tratement
weight | 8 week
  measure before and after tratement

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guthrie JR, Dennerstein L, Taffe JR, Donnelly V. Health care-seeking for menopausal problems. Climacteric. 2003 Jun;6(2):112-7. PMID 12841881
- See also: data obtain through the study may be provided to a qualified resarcher — https://www.who.int/news-room/fact-sheets/detail/menopause
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/12841881/